CLINICAL TRIAL: NCT04821414
Title: Effects of IL-1β and Its Receptor Antagonists in the Treatment of Severe Infection and Inflammatory Storm in Children
Status: Withdrawn | Type: Observational
Why Stopped: Lacking of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-19
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Critical Illness; Sepsis, Severe
Keywords: Critical Illness; Sepsis; anakinra; canakinumab; children
MeSH Terms: conditions — Critical Illness; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trial group: anakinra canakinumab
- control group: conventional treatment

SUMMARY:
In severe infective patients who survive the initial inflammatory storm, the immune response often evolves toward a state of immunosuppression, which contributes to increased mortality and severe secondary hospital-acquired infections. However, the role of IL-1β and its receptor antagonists in patients with severe sepsis and septic shock is discussed controversially. To date, the efficacy and safety of IL-1β and its receptor antagonists in children with severe infection is not fully evaluated.

DETAILED DESCRIPTION:
The investigators intend to enroll all children who were hospitalized in pediatric intensive care unit of Children's Hospital of Fudan University from January 2022 to December 2023. Children with a PICU length of day less than 48h will be excluded. Patients who met the inclusion criteria will be divided into trial group and control group. Clinical and demographic data, as well as treatment outcome will be collected from the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* Children between 29 days and 18 years old.
* Severe pneumonia and/or sepsis.
* Patients were included who meet the guideline for diagnosis and treatment of community-acquired pneumonia in Children (2019) issued by the National Health Commission of the people's Republic of China and/or who meet the International Guide to the 2020 campaign to Save sepsis: management of septic shock and sepsis-related organ dysfunction in children.

Exclusion Criteria:

* Notifiable infectious diseases.
* The researcher believes that he is not suitable to participate in other situations in this study.
* Participants in other clinical trials in the same period.
* Discharge within 48 hours

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children hospitalized in PICU of Children's Hospital of Fudan University from January 2022 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
survival rate | within 28 days after they discharged from PICU
  The death rate of children in 28 days after their discharged from PICU

SECONDARY OUTCOMES:
length of stay in PICU | within 28 days after they discharged from PICU
  Time from PICU admission to discharge